CLINICAL TRIAL: NCT06939686
Title: A Randomized Controlled Trial Evaluating Reprise Biomedical's Miro3D Wound Matrix and Standard of Care Versus Standard of Care Alone in Treating Wagner Grade 1 Diabetic Foot Ulcers and Dehiscence
Brief Title: Miro3D Wound Matrix Study for Diabetic Foot Ulcers and Wound Healing
Acronym: STRIDDDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reprise Biomedical, Inc. (Industry)
Collaborators: Barry University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REPRISE002; 20243362 (Other: WCG IRB)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcers (DFUs); Chronic Wound of the Lower Limb (Leg Ulcer or Foot Ulcer)
Keywords: Diabetic Foot Ulcer; Chronic Wound Healing; Miro3D Wound Matrix; Acellular Wound Scaffold; Porcine-derived Wound Matrix; Biologic Wound Matrix; Wound Granulation; Percentage Area Reduction; Reprise Biomedical
MeSH Terms: conditions — Diabetic Foot; Leg Ulcer; Foot Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Eligibility for Crossover: Subjects randomized to the SOC alone (control) arm who do not achieve complete healing of the index wound or ulcer by Week 12 are eligible to crossover into the Miro3D treatment phase.
  Crossover Treatment Plan:
  1. Subjects who opt into the crossover arm will begin treatment with Miro3D Wound Matrix plus SOC.
  2. Miro3D is applied weekly for the first 4 weeks.
  3. If the wound/ulcer remains unhealed after 4 weeks, application switches to biweekly (every 14 days).
  4. Treatment continues until healing is achieved or up to 12 weeks post-crossover, whichever comes first.
  Assessments During Crossover: Subjects are monitored weekly for:
  1. Percent Area Reduction (PAR)
  2. Granulation tissue formation
  3. Pain and Quality of Life (QOL) assessments
  4. Adverse Events (AEs) or Serious Adverse Events (SAEs)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Miro3D Wound Matrix plus Standard of Care (SOC) (Experimental): Subjects randomized to this arm receive Miro3D Wound Matrix in combination with standard of care wound treatment.
  * Miro3D is applied once every 7 days for the first 4 weeks.
  * If the wound is not healed after 4 weeks, Miro3D is applied biweekly (every 14 days) through week 12 or until healing.
  * All subjects in this arm are assessed weekly for healing progress, wound measurements, granulation, pain (VAS), and QOL.
  Interventions: Device: Miro3D Wound Matrix; Other: Standard of Care (SOC)
- Standard of Care (SOC) Alone (Active Comparator): Subjects in this arm receive standard wound care without Miro3D, including wound cleaning, debridement, offloading, and appropriate dressings.
  * Healing progress is evaluated weekly over the 12-week treatment period.
  * Subjects whose wounds remain unhealed at week 12 may elect to crossover to Miro3D treatment, following the same protocol used in Arm 1.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Device: Miro3D Wound Matrix — Miro3D is a sterile, acellular, three-dimensional biologic wound matrix derived from porcine liver via perfusion decellularization and drying. It is trimmed to fit the wound and rehydrated with sterile saline or Lactated Ringer's solution before application. It provides a porous scaffold to support granulation and healing in chronic or post-surgical wounds.
  Other Names: Miro3D
  Arms: Miro3D Wound Matrix plus Standard of Care (SOC)
Other: Standard of Care (SOC) — SOC includes standard wound care practices such as wound cleansing, debridement, infection management (if applicable), use of protective dressings (e.g., Aquacel or foam covered with Adaptic), and offloading devices (e.g., Foot Defender boot) to relieve pressure on the wound.
  Other Names: SOC

SUMMARY:
This study is a prospective, randomized controlled trial designed to evaluate the effectiveness of Miro3D Wound Matrix plus Standard of Care (SOC) compared to SOC alone in treating Wagner Grade 1 diabetic foot ulcers (DFUs) and wound dehiscence in an outpatient setting. The trial is sponsored by Reprise Biomedical, Inc. and aims to explore whether the addition of Miro3D-a three-dimensional, acellular porcine-derived wound matrix-enhances wound healing outcomes compared to SOC alone.

Purpose of the Study: The primary purpose of the study is to determine whether applying Miro3D in combination with SOC leads to improved healing of diabetic foot ulcers compared to SOC alone. Specifically, the study seeks to assess early wound healing progress at four weeks (as measured by percent area reduction and granulation tissue formation) as a predictor of complete healing by twelve weeks.

Key Question the Study Seeks to Answer: Does the addition of Miro3D to standard wound care improve the healing rate and overall wound outcomes for patients with Wagner Grade 1 diabetic foot ulcers or dehisced wounds compared to standard care alone?

Study Design Overview: Subjects who meet inclusion/exclusion criteria will be randomized into one of two groups:

1. Miro3D + SOC arm - receiving Miro3D weekly for 4 weeks, then biweekly if needed, for up to 12 weeks.
2. SOC alone (control) arm - receiving SOC without Miro3D. If the wound remains unhealed at 12 weeks in the SOC alone arm, participants may "crossover" to receive Miro3D treatment under the same schedule for an additional 12 weeks.

Primary Endpoint:

1. Percent Area Reduction (PAR) and granulation tissue formation at 4 weeks, serving as predictors for wound healing at 12 weeks.

Secondary Endpoints:

1. Quality of Life (QOL) improvements, including pain, mobility, and emotional well-being, assessed using a validated Wound/Ulcer-QOL tool.
2. Pain levels using a Visual Analog Scale (VAS) at each visit.

Population: Approximately 30 adult subjects (15 per arm) with Wagner Grade 1 diabetic foot ulcers or dehisced wounds will be enrolled. Subjects must have adequate blood flow, demonstrate wound size criteria, and commit to offloading and follow-up care.

Follow-Up: Subjects will be followed weekly through the 12-week study period. Healed subjects will undergo confirmation visits at 2 and 4 weeks post-closure. Subjects in the crossover arm will be followed for an additional 12 weeks if their wound was unhealed at the primary endpoint.

Statistical Considerations: Data will be summarized using descriptive statistics, including wound measurements, infection status, and healing rates. Comparative analysis will be conducted between treatment groups and schedules (weekly vs. biweekly Miro3D application). Adverse events (AEs), serious adverse events (SAEs), and device-related events will also be documented.

This study aims to generate clinical evidence supporting the use of Miro3D as a beneficial adjunct to standard wound care in promoting early and complete healing of diabetic foot ulcers.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial evaluates the clinical effectiveness of Reprise Biomedical's Miro3D Wound Matrix in conjunction with standard of care (SOC) compared to SOC alone in treating Wagner Grade 1 diabetic foot ulcers (DFUs) in an outpatient setting. The investigational product, Miro3D, is a porcine liver-derived, acellular, three-dimensional extracellular matrix designed to support healing in complex wound environments by providing a biologically active scaffold that facilitates cell infiltration and tissue remodeling. This study aims to generate robust clinical evidence supporting Miro3D's role as an advanced biologic dressing for early and sustained wound healing in diabetic patients.

Background and Rationale: Diabetic foot ulcers are a common and serious complication of diabetes mellitus, affecting approximately 15-25% of individuals with diabetes over their lifetime. These ulcers are associated with high morbidity, increased healthcare utilization, and significant risk of lower extremity amputation. Despite established guidelines, many DFUs fail to heal adequately with standard of care alone, especially when early progress is not observed. According to consensus recommendations, wounds that do not demonstrate at least a 50% reduction in area within the first four weeks of SOC are unlikely to achieve closure by 12 weeks and are considered candidates for advanced wound therapies.

Advanced biologic matrices aim to address the limitations of SOC by enhancing the local wound environment. Miro3D is a perfusion-decellularized extracellular matrix derived from porcine liver, preserving native microvascular architecture and providing a highly porous scaffold for cellular infiltration. Unlike many sheet-based dermal matrices, Miro3D possesses significant three-dimensional structure and volume, making it suitable for filling shallow to moderately deep wound beds. The device is supplied sterile and dry, rehydrated at the point of care, trimmed to fit, and applied directly to the wound bed.

This study is designed to evaluate whether the addition of Miro3D to SOC accelerates healing and improves outcomes in Wagner Grade 1 DFUs, a common clinical presentation that often remains refractory to SOC alone. The trial also includes a crossover design for non-responders in the SOC arm, enhancing ethical treatment access while generating additional observational data.

Device Description and Mechanism of Action: Miro3D Wound Matrix is a sterile, acellular scaffold composed of porcine-derived extracellular matrix processed via perfusion decellularization to retain native liver architecture. The matrix is characterized by high porosity, preserved vascular pathways, and structural integrity, supporting rapid integration into the wound bed. Once rehydrated, Miro3D becomes pliable and conformable, suitable for application to irregular wound geometries.

Mechanistically, Miro3D provides a physical and biochemical scaffold that promotes cell adhesion, migration, angiogenesis, and granulation. As a non-crosslinked, resorbable collagen matrix, it undergoes host remodeling over time, integrating into newly formed tissue. The device can be trimmed to wound dimensions and applied weekly or biweekly depending on healing progression.

Study Objectives and Hypothesis: The primary objective of the study is to determine whether the application of Miro3D in combination with SOC leads to superior healing outcomes compared to SOC alone in the treatment of Wagner Grade 1 DFUs.

Primary Hypothesis: Miro3D + SOC will result in a significantly higher proportion of wounds achieving ≥50% area reduction and robust granulation tissue formation at 4 weeks, predictive of complete closure by 12 weeks.

Secondary Hypotheses: Subjects treated with Miro3D + SOC will demonstrate faster time to healing, improved patient-reported quality of life (QOL), reduced pain, and comparable or improved safety compared to those receiving SOC alone.

Study Design and Randomization: This is a randomized controlled trial enrolling approximately 30 subjects (15 per arm). Subjects meeting eligibility criteria will be randomized in a 1:1 ratio to either:

1. Intervention Arm (Miro3D + SOC): Weekly Miro3D application for the first four weeks, followed by biweekly application if the wound remains unhealed, for up to 12 weeks.
2. Control Arm (SOC alone): Standard wound care practices without Miro3D. Subjects with unhealed wounds at 12 weeks are eligible to cross over to receive Miro3D under the same application schedule for an additional 12-week observational phase.

Randomization will use sealed envelope assignment to ensure unbiased group assignment.

Visit Schedule and Study Assessments:

1. Screening Visit (Week -2 to 0):

   * Informed consent
   * Wound debridement and imaging
   * Vascular assessment
   * HbA1c testing, pregnancy test if applicable
   * Run-in period
2. Randomization Visit (Week 0):

   * Confirm eligibility
   * Randomization
   * Baseline wound measurements and photos
   * QOL and pain scale assessments
   * First application of Miro3D (intervention arm)
3. Weekly Treatment Visits (Weeks 1-11):

   * Wound imaging and measurements
   * Clinical assessment and re-debridement as needed
   * Miro3D reapplication (as indicated)
   * Pain assessment and adverse event tracking
4. End-of-Treatment Visit (Week 12):

   * Final wound assessment
   * Confirmation of wound closure
   * Final QOL and pain scale assessments
   * Eligibility for crossover (control arm, if unhealed)
5. Crossover Phase (Weeks 13-24, as needed):

   * Subjects from SOC arm receive Miro3D + SOC
   * Follow-up per the intervention arm protocol
6. Closure Confirmation Visits (2 and 4 weeks post-closure):

   * Validation of sustained healing

Crossover Design and Follow-Up: Subjects in the SOC arm who do not achieve complete healing by Week 12 are eligible to cross over to receive Miro3D under the same application schedule. The crossover phase is observational and not included in the primary efficacy analysis. These data will help characterize Miro3D's performance as a rescue therapy in chronic wounds unresponsive to SOC.

Subjects who achieve healing during the randomized phase or crossover phase will undergo 2- and 4-week confirmation visits to validate sustained closure.

Safety Monitoring and Adverse Event Reporting: All adverse events will be documented, assessed for severity and relatedness, and reported per FDA and IRB requirements. Investigators will monitor subjects for infection, delayed healing, inflammatory reactions, and systemic complications. Device-related events will be tracked by lot number.

Unanticipated adverse device effects (UADEs), if any, will be escalated to the sponsor and appropriate regulatory bodies. Based on previous clinical use of hepatic-derived ECM scaffolds, Miro3D is expected to demonstrate a favorable safety profile.

Regulatory, Ethical, and Clinical Context: Miro3D Wound Matrix is FDA-cleared under 510(k) as a Class II medical device (K223257) for use in managing partial- and full-thickness wounds. This trial is conducted as a post-market, investigator-initiated study in accordance with Good Clinical Practice (GCP), IRB approval, and informed consent regulations under 21 CFR Part 50.

The trial addresses a critical gap in clinical evidence by comparing Miro3D to SOC in a randomized, controlled framework. Few biologic wound matrices have RCT-level data supporting early use in Wagner Grade 1 DFUs. The findings will inform clinical guidelines, payer coverage decisions, and the design of larger-scale trials aimed at improving outcomes for patients with chronic diabetic wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age and capable of providing informed consent.
2. Must have a full- or partial-thickness Wagner Grade 1 ulcer or wound on the foot; if involving the malleolus, no more than 50% of the wound may be above the midpoint of the medial malleolus.
3. Index wound/ulcer must be between 1 cm² and 20 cm² post-debridement.
4. Wound/ulcer must have been present for at least 4 weeks prior to screening.
5. Adequate circulation must be documented by one of the following: ABI between 0.7-1.2, TBI ≥ 0.7, TCPO2 ≥ 40 mmHg, or triphasic/biphasic Doppler waveforms.
6. Other wounds, if present, must be at least 2 cm from the index wound/ulcer.
7. Any previous infections must have been adequately treated per IDSA guidelines.
8. Subjects must agree to proper offloading and/or compression, have a stable living environment, and be able to attend follow-up visits.
9. Must provide written consent for digital imaging.
10. For Miro3D arm: Index wound/ulcer must have a clean base free of devitalized tissue or debris at the time of product placement.

Exclusion Criteria:

1. Index wound/ulcer has reduced ≥30% after two weeks of SOC from screening to baseline.
2. Poorly controlled diabetes (HbA1c ≥ 12%).
3. Active, untreated or uncontrolled osteomyelitis.
4. Malignancy or vasculitis at the wound site.
5. Undergoing chemotherapy.
6. On dialysis.
7. Use of investigational drugs or therapies within 30 days prior to screening.
8. Conditions that would compromise study participation or adherence.
9. Known sensitivity to porcine materials.
10. Third-degree burns.
11. Worsening ischemia or gangrene at screening.
12. History of radiation to the wound site.
13. Exposed internal fixation, implants, or hardware in the wound.
14. Patient is transitioning to palliative or comfort care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Percent Area Reduction (PAR) and Granulation Tissue Formation at 4 Weeks | 4 weeks post-randomization
  The primary endpoint is the percent area reduction (PAR) and granulation tissue formation of the index wound or ulcer measured at 4 weeks. This serves as a predictor of complete healing by week 12. Wound size is measured manually using a ruler, and depth is assessed with a probe. Granulation is visually assessed by trained clinicians.

SECONDARY OUTCOMES:
Complete Wound or Ulcer Healing by Week 12 | Up to 12 weeks post-randomization
  The proportion of subjects whose index wound or ulcer is fully healed (defined as full epithelialization without drainage) at or before week 12. Closure must be sustained for 4 consecutive weeks and confirmed by follow-up visits.
Quality of Life (QOL) Assessment Using Wound-QOL Instrument | Baseline, Week 4, Week 8, and Week 12 or at early termination
  Change from baseline in subject-reported quality of life using the Wound-QOL tool, which assesses domains such as pain, odor, physical function, mobility, depression, and social isolation.
Pain Score Assessment Using Visual Analog Scale (VAS) | Collected at every study visit (weekly through week 12)
  Change from baseline in pain intensity as measured by a standard 0-10 Visual Analog Scale (VAS), where 0 represents no pain and 10 represents worst possible pain.

OTHER OUTCOMES:
Healing Trajectory at Weeks 6 and 8 | 6 weeks and 8 weeks post-randomization
  Interim assessments of percent area reduction (PAR) and granulation at weeks 6 and 8 to evaluate healing trajectory and likelihood of closure by week 12.
Safety Profile: Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Device Effects (UADEs) | From informed consent through 30 days post-final study visit
  Collection and evaluation of all adverse events, serious adverse events, and unanticipated adverse device effects. Events will be assessed for severity, expectedness, and relationship to the study device or SOC.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Snyder, DPM, Principal Investigator — Barry University
Locations (3):
- United States (3):
  - West Boca Center for Wound Healing, Coconut Creek, Florida
  - Barry University Clinical Research, Tamarac, Florida
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warriner RA, Snyder RJ, Cardinal MH. Differentiating diabetic foot ulcers that are unlikely to heal by 12 weeks following achieving 50% percent area reduction at 4 weeks. Int Wound J. 2011 Dec;8(6):632-7. doi: 10.1111/j.1742-481X.2011.00860.x. Epub 2011 Sep 23. PMID 21951763
- [Background] Snyder RJ, Cardinal M, Dauphinee DM, Stavosky J. A post-hoc analysis of reduction in diabetic foot ulcer size at 4 weeks as a predictor of healing by 12 weeks. Ostomy Wound Manage. 2010 Mar 1;56(3):44-50. PMID 20368673
- [Background] Smith ME, Totten A, Hickam DH, Fu R, Wasson N, Rahman B, Motu'apuaka M, Saha S. Pressure ulcer treatment strategies: a systematic comparative effectiveness review. Ann Intern Med. 2013 Jul 2;159(1):39-50. doi: 10.7326/0003-4819-159-1-201307020-00007. PMID 23817703
- [Background] Raghav A, Khan ZA, Labala RK, Ahmad J, Noor S, Mishra BK. Financial burden of diabetic foot ulcers to world: a progressive topic to discuss always. Ther Adv Endocrinol Metab. 2018 Jan;9(1):29-31. doi: 10.1177/2042018817744513. Epub 2017 Dec 12. PMID 29344337
- [Background] Padula WV, Delarmente BA. The national cost of hospital-acquired pressure injuries in the United States. Int Wound J. 2019 Jun;16(3):634-640. doi: 10.1111/iwj.13071. Epub 2019 Jan 28. PMID 30693644
- [Background] Mervis JS, Phillips TJ. Pressure ulcers: Pathophysiology, epidemiology, risk factors, and presentation. J Am Acad Dermatol. 2019 Oct;81(4):881-890. doi: 10.1016/j.jaad.2018.12.069. Epub 2019 Jan 18. PMID 30664905
- [Background] Kruger EA, Pires M, Ngann Y, Sterling M, Rubayi S. Comprehensive management of pressure ulcers in spinal cord injury: current concepts and future trends. J Spinal Cord Med. 2013 Nov;36(6):572-85. doi: 10.1179/2045772313Y.0000000093. Epub 2013 May 21. PMID 24090179
- [Background] Geriatric Medicine Gerontology Chapter 30 - Pressure Ulcers. (n.d.). Retrieved from Johns Hopkins: https://www.hopkinsmedicine.org/geriatric_medicine_gerontology/_downloads/readings/section8.pdf
- [Background] Bauer K, Rock K, Nazzal M, Jones O, Qu W. Pressure Ulcers in the United States' Inpatient Population From 2008 to 2012: Results of a Retrospective Nationwide Study. Ostomy Wound Manage. 2016 Nov;62(11):30-38. PMID 27861135
- See also: Miro3D Wound Matrix product webpage — https://reprisebio.com/miro3d/